CLINICAL TRIAL: NCT02905370
Title: Progressing Home Health Rehabilitation Paradigms for Older Adults
Brief Title: Progressing Home Health Rehabilitation for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Arcadia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-2125; R01NR016209 (NIH)
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Older Adults; Physical Deconditioning
Keywords: Home Health; Rehabilitation; High Intensity; Hospital Associated Deconditioning; Functional Mobility; Physical Function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Progressive Multi-Component (PMC) (Experimental): High intensity strength training protocol, daily protein supplementation, functionally enhanced transitions of care
  Interventions: Behavioral: Progressive Multi-Component (PMC)
- Enhanced Usual Care (EUC) (Active Comparator): Low intensity rehabilitation protocol, standard education for nutrition, standard transitions of care
  Name of Participant Arm updated to "Enhanced Usual Care" from "Usual Care" effective 8/16/18 to distinguish from Passive Comparator "True Usual Care" group.
  Interventions: Behavioral: Enhanced Usual Care (EUC)
- True Usual Care (TUC) (No Intervention): Real-world home health rehabilitation, real-world education for nutrition, real-world transitions of care, non-randomized observation
  Participants in the "True Usual Care" group will receive physical therapy following discharge from acute hospitalization. Activities and number of visits are not protocolized and are provided by real world home health care providers per physician orders.
  Participant Arm added effective 8/16/18.

INTERVENTIONS:
Behavioral: Progressive Multi-Component (PMC) — Participants in the "Progressive Multi-component" intervention group will receive 1) high intensity physical therapy, 2) protein supplement, and 3) emphasis on functionally enhanced transitions of care following discharge from post-acute setting. High intensity physical therapy will include progressive resistance training, multi-planar motor control and gait exercises, and high intensity activities of daily living training. Functionally enhanced transitions of care protocol includes a personal health record with 5 domains that are addressed in an interdisciplinary manner with the patient. Participants will receive 12 intervention visits over 60 days. Participants will also receive a home exercise program.
  Arms: Progressive Multi-Component (PMC)
Behavioral: Enhanced Usual Care (EUC) — Participants in the "Enhanced Usual Care" group will receive standardized physical therapy following discharge from acute hospitalization. The activities of therapy will include basic strength training, single-planar motor control and gait exercises, and activities of daily living training. Participants will receive 12 intervention visits over 60 days. Participants will also receive a standardized home exercise program and standard nutritional education.
  Name of Participant Arm updated to "Enhanced Usual Care" from "Usual Care" effective 8/16/18 to distinguish from Passive Comparator "True Usual Care" group.
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
This research study explores the effects of a progressive, multi-component intervention following a stay in the hospital or rehabilitation facility. The purpose of this research study is to compare a multi-component intervention (higher intensity exercise, nutritional supplementation, and greater emphasis on functionally enhanced care transitions) with usual care physical therapy.

DETAILED DESCRIPTION:
Declines in physical function as a result of acute illness are strongly and independently associated with a number of adverse health events for older adults. Home Health (HH) physical therapy may be the ideal venue for addressing these declines in physical function because around 3 million older adults receive HH services following discharge from acute or post-acute facilities. However, as currently structured, HH care does not appear to adequately restore function, as evidenced by poor long-term outcomes and high rates of hospital readmission. Diminished physical function has been particularly implicated as a risk factor for re-hospitalization --older adults with lower levels of ambulatory activity are 6 times more likely to be re-hospitalized than those with greater ambulatory activity. A more intensive approach to HH physical therapy for older adults has great potential to maximize physical function and reduce hospital readmissions. Therefore, the investigators have developed a high intensity home-based, progressive, interdisciplinary, multi-component (PMC) intervention that directly addresses the functional deficits seen after hospitalization. This intervention will include intensive rehabilitation, a care transitions program, and daily protein supplementation. The investigators will conduct a two-arm, randomized clinical trial (RCT) of 200 participants admitted to HH from an acute or post-acute facility. Participants will receive either 1) an intensive, PMC intervention using resistance exercise and evidenced-based motor control training to improve physical function, along with nutritional supplementation and emphasis on functionally enhanced care transitions or 2) usual care (UC) physical therapy. The primary goal of this investigation is to determine if PMC intervention, initiated upon admission to HH, improves physical function, as measured by performance and self-report assessments, more than UC physical therapy. The investigators will also examine the effects on fatigue, balance confidence, and activities of daily living. In an exploratory analysis, the effects of the PMC intervention on re-hospitalization rates, nursing home placement, emergency room visits, and falls after discharge from the acute care hospital will also be examined. All outcomes will be examined at baseline, 30, 60 (primary endpoint), 90 and 180 days. If successful in improving patient function and decreasing re-hospitalization rates, PMC intervention holds potential for future health care cost savings.

ELIGIBILITY:
Inclusion Criteria:

1. 65 years of age and older
2. Referred to home care physical therapy following acute medical deconditioning
3. Have at least 3 comorbid conditions including those listed below:

   * Chronic Obstructive Pulmonary Disease
   * Gastrointestinal Bleed
   * Urinary Tract Infection
   * Pneumonia
   * Chronic ulcerative wounds
   * Diabetes
   * Hypertension
   * Depression/mental health
   * Irritable Bowel Syndrome
   * Hernia
   * Post-op pancreatic surgery
   * Osteoporosis/OA/RA/Gout
   * Heart Disease
   * Hypercholesterolemia
   * Peripheral Arterial Disease
   * Spinal Stenosis
   * Dehydration
   * Syncope
   * Atrial fibrillation
   * Hypo/Hyperthyroid
   * Renal Failure (no dialysis)
   * Post-op bowel surgery
   * Congestive Heart Failure
4. Be ambulatory without human assistance prior to hospitalization
5. Be English-speaking

Exclusion Criteria: (one or more):

1. Acute lower extremity fracture with weight-bearing restriction
2. "Elective" joint replacement surgery
3. Lower extremity amputation
4. Acute cardiac surgery
5. Terminal illness
6. Active cancer treatment in which exercise is contraindicated
7. Deep vein thrombosis/pulmonary embolus (DVT/PE)
8. Recent stroke (within 1 yr)
9. Score of <20 on SLUMS (as of 08.16.2018, revised to exclusion #14)
10. Inability to ambulate 10 feet without human assistance at time of hospital discharge
11. Gait Speed <0.3m/s or >1.0 m/s
12. Progressive neurodegenerative diagnosis (e.g. Parkinson's, MS, ALS)
13. Use of illegal substances
14. Clinical discretion of study physician to exclude patients who are determined to be unsafe and/or inappropriate to participate in high intensity rehabilitation as defined by the inclusion/exclusion criteria
15. Active involvement of Adult Protection Services
16. Current dialysis treatment
17. Prisoners or those on probation or other alternative sentencing

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 353 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2022-05-06 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Short Physical Performance Battery (SPPB) | Change in SPPB from baseline to 60 days post randomization
  SPPB is a well-accepted global measure of lower extremity function which consists of walking speed, chair stands, and balance. It is a well-studied composite measure and a strong predictor of disability, institutionalization, and morbidity in older adults. SPPB will also be assessed at 30, 90, 180 days post-randomization.

SECONDARY OUTCOMES:
Modified Physical Performance Test (mPPT) | Change in mPPT from baseline to 60 days post randomization
  mPPT assesses 7 tasks. Based on the time it takes to complete each task, a score from 0 (unable to complete) to 4 (performed quickly and easily) is given for each item. The maximal score is 28 and includes tasks that involve upper and lower extremity function. Test-retest reliability for the modified PPT score is 0.96. The instrument is sensitive to change and has been used in exercise trials with frail elders. mPPT will also be assessed at 30, 90, 180 days post-randomization.
Fast walking speed (4MW) | Change in 4MW from baseline to 60 days post randomization
  Will be assessed at the fastest, safe speed for each participant over 4 meters. Fastest walking assesses capacity for performance of certain activities (e.g. crossing a street before the light changes). Fast walking speed will also be assessed at 30, 90, 180 days post-randomization.
ActivPAL | Change in physical activity from baseline to 60 days post randomization
  Accelerometer-based physical activity examines volume and intensity of physical activity in which participants engage. Participants will wear a thigh-mounted activPAL physical activity monitoring device for up to 10 days to determine mean steps and activity counts per day (PAL Technologies, Glasgow, Scotland). Physical activity will also be defined as daily time spent in sitting, standing, and stepping. The activPAL has been found to be reliable (ICC≥0.99), valid (% Error =0.94% compared to video analysis; gold standard), and suitably sensitive to detect difference/change is similar populations. Physical activity will also be assessed at 30, 90, 180 days post-randomization.
Falls Efficacy Scale-International | Change in Falls Efficacy Scale-International from baseline to 60 days post randomization
  Questionnaire assesses concern about falling during performance of activities of daily living. Participants rate 16 individual activities on a scale from 1 (not at all concerned) to 4 (very concerned). Falls Efficacy Scale-International will also be assessed at 30, 90, 180 days post-randomization.
Fatigue Severity Scale (FSS) | Change in FSS from baseline to 60 days post randomization
  A nine item questionnaire that quantifies the degree of fatigue and the impact of fatigue on activities of daily living in clinical populations. Participants score each of 9 components on a scale of 1 to 7. The aggregate score ranges from 9 (no impact) to 64 (profound impact of fatigue on activities of daily living). A total score of less than 36 suggests that a participant is not suffering from fatigue. The FSS is reliable (r=0.56-0.89), valid (α=0.97), and sensitive to change. FSS will also be assessed at 30, 90, 180 days post-randomization.
Patient Activation Measure (PAM) | Change in PAM from baseline to 60 days post randomization
  Identifies patient motivation levels regarding their healthcare. Reliably predicts future ER visits, hospital admissions, and medication/ therapy adherence. The survey classifies patient activation levels on a scale from 1 (low activation/motivation) to 4 (high activation/motivation). Patients who score higher on the PAM survey tend to be hospitalized less and adhere to medication and therapy schedules more.
Grip Strength | Change in Grip Strength from baseline to 60 days post randomization
  Grip strength is a simple and reliable surrogate of overall muscle strength and a valid predictor of physical disability and mobility limitation. Grip strength will also be assessed at 30, 90, 180 days post-randomization.

OTHER OUTCOMES:
Falls, Emergency Department visits, nursing home days, hospitalizations | Quantification of falls, ED visits, nursing home days, and hospitalizations at 30, 60, 90, and 180 days post randomization
  Patients will be given a log to record any falls, ED visits, hospitalizations or nursing home stays. Falls will be defined as an unintentional change in position resulting in coming to rest on the ground or other lower level.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer E Stevens-Lapsley, MPT, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver, Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cawood AL, Elia M, Stratton RJ. Systematic review and meta-analysis of the effects of high protein oral nutritional supplements. Ageing Res Rev. 2012 Apr;11(2):278-96. doi: 10.1016/j.arr.2011.12.008. Epub 2011 Dec 22. PMID 22212388
- [Background] Fisher SR, Kuo YF, Sharma G, Raji MA, Kumar A, Goodwin JS, Ostir GV, Ottenbacher KJ. Mobility after hospital discharge as a marker for 30-day readmission. J Gerontol A Biol Sci Med Sci. 2013 Jul;68(7):805-10. doi: 10.1093/gerona/gls252. Epub 2012 Dec 19. PMID 23254776
- [Background] Murkofsky RL, Alston K. The past, present, and future of skilled home health agency care. Clin Geriatr Med. 2009 Feb;25(1):1-17, v. doi: 10.1016/j.cger.2008.11.006. PMID 19217489
- [Background] Solomon DH, Wagner DR, Marenberg ME, Acampora D, Cooney LM Jr, Inouye SK. Predictors of formal home health care use in elderly patients after hospitalization. J Am Geriatr Soc. 1993 Sep;41(9):961-6. doi: 10.1111/j.1532-5415.1993.tb06762.x. PMID 8409182
- [Background] Timmer AJ, Unsworth CA, Taylor NF. Rehabilitation interventions with deconditioned older adults following an acute hospital admission: a systematic review. Clin Rehabil. 2014 Nov;28(11):1078-86. doi: 10.1177/0269215514530998. Epub 2014 May 20. PMID 24844238
- [Derived] Falvey JR, Mangione KK, Nordon-Craft A, Cumbler E, Burrows KL, Forster JE, Stevens-Lapsley JE. Progressive Multicomponent Intervention for Older Adults in Home Health Settings Following Acute Hospitalization: Randomized Clinical Trial Protocol. Phys Ther. 2019 Sep 1;99(9):1141-1149. doi: 10.1093/ptj/pzz069. PMID 31004493

DOCUMENTS (4):
  • Informed Consent Form: Consent (2021-09-17): https://cdn.clinicaltrials.gov/large-docs/70/NCT02905370/ICF_000.pdf
  • Informed Consent Form: Consent SOC (2021-09-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT02905370/ICF_001.pdf
  • Informed Consent Form: VA Consent (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT02905370/ICF_002.pdf
  • Informed Consent Form: VA Consent SOC (2021-12-08): https://cdn.clinicaltrials.gov/large-docs/70/NCT02905370/ICF_003.pdf